CLINICAL TRIAL: NCT03844880
Title: Emotional Awareness and Expression Therapy (EAET) or Cognitive Behavior Therapy (CBT) for the Treatment of Chronic Musculoskeletal Pain in Older Veterans: A Pilot Randomized Clinical Trial
Brief Title: Emotional Awareness and Expression Therapy (EAET) or Cognitive Behavior Therapy (CBT) for Older Veterans With Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2018-12-19; First posted 2019-02-19 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic Pain; Psychotherapy; Musculoskeletal Disease
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Musculoskeletal Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Awareness and Expression Therapy (Experimental): Seeks to reduce physical (e.g., pain) and emotional (e.g., depression, anxiety) symptoms by helping individuals become aware of their emotions, express them, and resolve emotional conflicts. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy
- Cognitive Behavior Therapy (Active Comparator): Seeks to help individuals function better and improve symptoms by teaching various cognitive and behavioral skills to manage symptoms. It will use techniques such as relaxation training, engaging in pleasant activities, pacing yourself, and changing unhelpful ways of thinking.
  Interventions: Behavioral: Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — Focus on emotions, writing about stress, assertiveness training, role playing new ways to handle relationships, and sharing feelings and experiences with others.
  Arms: Emotional Awareness and Expression Therapy
Behavioral: Cognitive Behavior Therapy — Focus on cognitive and behavioral skills, such as relaxation, increasing pleasant activities, pacing, and changing ways of thinking.
  Arms: Cognitive Behavior Therapy

SUMMARY:
A randomized clinical trial for Veterans age 50 years and older with chronic musculoskeletal pain in which Emotional Awareness and Expression Therapy (EAET) is compared against Cognitive Behavior Therapy (CBT) to evaluate acceptability, feasibility, and efficacy of the two treatments on pain and other outcomes, as well as potential mediators of treatment response.

DETAILED DESCRIPTION:
Outpatient Veterans age 50 years and older at the West Los Angeles VA Medical Center who have chronic musculoskeletal pain complete baseline questionnaires and are randomized into one of two forms of psychotherapy: Emotional Awareness and Expression Therapy (EAET), which helps patients make connections between avoided or conflicted emotions and pain, or Cognitive Behavior Therapy (CBT), which teaches pain coping skills. Each treatment is delivered by an experienced therapist and includes one 90-minute individual session and eight 90-minute group sessions (in small groups of 8 Veterans). Patients in both conditions complete post-treatment and 3-month follow-up questionnaires. Outcomes of each type of psychotherapy are compared and mediators of treatment response are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Veteran;
* Age 50 years and older;
* 3 months of musculoskeletal pain including low back pain and other regional pain syndromes (e.g. neck, leg, pelvic pain and temporomandibular joint disorders), whiplash, widespread pain (e.g. fibromyalgia), or tension headaches.

Exclusion Criteria:

* Leg pain greater than back pain (to exclude radiculopathy in isolation);
* Electromyography (EMG)-confirmed "tunnel" syndromes (e.g. carpal or tarsal tunnel syndrome) without any other pain complaints;
* Autoimmune disease that typically generates pain (e.g. systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, ankylosing spondylitis);
* Confirmed hip or knee osteoarthritis without any other pain complaints;
* Cancer pain, sickle cell disease, neuralgias (e.g. trigeminal neuralgia), burn pain, infection associated with pain (e.g. vertebral infection), cauda equina syndrome, gout as the only pain complaint, migraine or cluster headaches only;
* Uncontrolled severe psychiatric disorder including current psychotic disorder (e.g. schizophrenia or bipolar I disorder not controlled with medications), dissociative identity disorder, or active suicide/violence risk in the past 6 months;
* Moderate to severe cognitive impairment or dementia (Mini-Mental State Exam score ≤ 25);
* Active severe alcohol or substance use disorder that inhibits the participant's ability to attend sessions or participate in homework;
* Currently with pain-related litigation or applying for compensation or compensation increase (e.g. applying for VA service connection or applying for VA service connection increase for pain);
* Unable to fluently read/converse in English;
* Planning to move from the area in the next 6 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Mean Pain Severity | Change from baseline to 8 weeks
  Average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10.
Mean Pain Severity | Change from baseline to 20 weeks
  Average of 4 self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be), yielding a total score between 0 and 10.

SECONDARY OUTCOMES:
Percent of Group Therapy Sessions Attended | 8 weeks
  Number of sessions each participant attends divided by 8 sessions (total number of sessions available to attend).
Satisfaction with Therapy and Therapist Scale-Revised | 8 weeks
  Satisfaction with therapy subscale is the summation of 6 items, each scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction), yielding a total score between 6 and 30. Satisfaction with therapist subscale is the summation of 6 items, each scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction), yielding a total score between 6 and 30. Overall satisfaction is an additional single item scored 1-5 (1 = maximum dissatisfaction; 5 = maximum satisfaction). The two subscales and the overall satisfaction item are each reported separately.
Patient Reported Outcomes Measurement Information System (PROMIS)-Pain Behavior Short Form 7a v1.1 | Change from baseline to 8 weeks
  Sum of seven self-report items assessing behaviors associated with pain over the past 7 days. Items range from 1-6 (1 = had no pain; 6 = always), yielding a total score between 7 and 42.
PROMIS-Pain Behavior Short Form 7a v1.1 | Change from baseline to 20 weeks
  Sum of seven self-report items assessing behaviors associated with pain over the past 7 days. Items range from 1-6 (1 = had no pain; 6 = always), yielding a total score between 7 and 42.
PROMIS-Pain Interference Short Form 8a v1.0 | Change from baseline to 8 weeks
  Sum of eight self-report items assessing interference of pain with daily activities over the past 7 days. Items range from 1-5 (1 = no interference; 5 = maximum interference), yielding a total score between 8 and 40.
PROMIS-Pain Interference Short Form 8a v1.0 | Change from baseline to 20 weeks
  Sum of eight self-report items assessing interference of pain with daily activities over the past 7 days. Items range from 1-5 (1 = no interference; 5 = maximum interference), yielding a total score between 8 and 40.
PROMIS-Depression Short Form | Change from baseline to 8 weeks
  Sum of eight self-report items assessing depression and emotional distress over the past 7 days. Items range from 1-5 (1 = never feeling a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 8 and 40.
PROMIS-Depression Short Form | Change from baseline to 20 weeks
  Sum of eight self-report items assessing depression and emotional distress over the past 7 days. Items range from 1-5 (1 = never feeling a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 8 and 40.
PROMIS-Anxiety Short Form | Change from baseline to 8 weeks
  Sum of seven self-report items assessing anxiety over the past 7 days. Items range from 1-5 (1 = never experiencing a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 7 and 35.
PROMIS-Anxiety Short Form | Change from baseline to 20 weeks
  Sum of seven self-report items assessing anxiety over the past 7 days. Items range from 1-5 (1 = never experiencing a type of distressing emotion; 5 = always feeling that emotion), yielding a total score between 7 and 35.
PTSD Symptom Scale | Change from baseline to 8 weeks
  Sum of seventeen self-report items assessing PTSD according to the frequency in which symptoms are experienced over the last two weeks. Items range from 0-3 (0 = not experiencing a symptom; 1 = once per week or less / a little bit / once in a while; 2 = 2 to 4 times per week / somewhat / half the time; 3 = 3 to 5 or more times per week / very much / almost always), yielding a total score between 0 and 51.
PTSD Symptom Scale | Change from baseline to 20 weeks
  Sum of seventeen self-report items assessing PTSD according to the frequency in which symptoms are experienced over the last two weeks. Items range from 0-3 (0 = not experiencing a symptom; 1 = once per week or less / a little bit / once in a while; 2 = 2 to 4 times per week / somewhat / half the time; 3 = 3 to 5 or more times per week / very much / almost always), yielding a total score between 0 and 51.
NIH Toolbox-Positive Affect Short Form | Change from baseline to 8 weeks
  Sum of fifteen self-report items assessing positive affect over the past 7 days. Items range from 1-5 (1 = not at all experiencing a type of positive emotion; 5 = very much feeling that emotion), yielding a total score between 15 and 75.
NIH Toolbox-Positive Affect Short Form | Change from baseline to 20 weeks
  Sum of fifteen self-report items assessing positive affect over the past 7 days. Items range from 1-5 (1 = not at all experiencing a type of positive emotion; 5 = very much feeling that emotion), yielding a total score between 15 and 75.
NIH Toolbox-Purpose and Meaning Short Form | Change from baseline to 8 weeks
  Sum of seven self-report items assessing general feelings of meaning and purpose. Items range from 1-5 (1 = no purpose and meaning; 5 = maximum purpose and meaning), yielding a total score between 7 and 35.
NIH Toolbox-Purpose and Meaning Short Form | Change from baseline to 20 weeks
  Sum of seven self-report items assessing general feelings of meaning and purpose. Items range from 1-5 (1 = no purpose and meaning; 5 = maximum purpose and meaning), yielding a total score between 7 and 35.
NIH Toolbox-Life Satisfaction Short Form | Change from baseline to 8 weeks
  Sum of five self-report items assessing general life satisfaction. Items range from 1-5 (1 = no satisfaction; 5 = maximum satisfaction), yielding a total score between 5 and 25.
NIH Toolbox-Life Satisfaction Short Form | Change from baseline to 20 weeks
  Sum of five self-report items assessing general life satisfaction. Items range from 1-5 (1 = no satisfaction; 5 = maximum satisfaction), yielding a total score between 5 and 25.
PROMIS-Sleep Disturbance Short Form | Change from baseline to 8 weeks
  Sum of eight self-report items assessing sleep disturbance over the past 7 days. Items range from 1-5 (1 = no sleep disturbance; 5 = maximum sleep disturbance), yielding a total score between 8 and 40.
PROMIS-Sleep Disturbance Short Form | Change from baseline to 20 weeks
  Sum of eight self-report items assessing sleep disturbance over the past 7 days. Items range from 1-5 (1 = no sleep disturbance; 5 = maximum sleep disturbance), yielding a total score between 8 and 40.
PROMIS-Fatigue Short Form | Change from baseline to 8 weeks
  Sum of seven self-report items assessing fatigue over the past 7 days. Items range from 1-5 (1 = no fatigue; 5 = maximum fatigue), yielding a total score between 7 and 35.
PROMIS-Fatigue Short Form | Change from baseline to 20 weeks
  Sum of seven self-report items assessing fatigue over the past 7 days. Items range from 1-5 (1 = no fatigue; 5 = maximum fatigue), yielding a total score between 7 and 35.
Multidimensional Inventory of Subjective Cognitive Impairment | Change from baseline to 8 weeks
  Sum of ten self-report items assessing subjective cognitive impairment over the past 7 days. Items range from 1-5 (1 = no impairment; 5 = maximum impairment), yielding a total score between 10 and 50.
Multidimensional Inventory of Subjective Cognitive Impairment | Change from baseline to 20 weeks
  Sum of ten self-report items assessing subjective cognitive impairment over the past 7 days. Items range from 1-5 (1 = no impairment; 5 = maximum impairment), yielding a total score between 10 and 50.
Ambivalence over Emotional Expression Questionnaire | Change from baseline to 8 weeks
  Sum of fourteen self-report items assessing ambivalence of emotional expression. Items range from 1-5 (1 = no ambivalence; 5 = maximum ambivalence), yielding a total score between 14 and 70.
Ambivalence over Emotional Expression Questionnaire | Change from baseline to 20 weeks
  Sum of fourteen self-report items assessing ambivalence of emotional expression. Items range from 1-5 (1 = no ambivalence; 5 = maximum ambivalence), yielding a total score between 14 and 70.
Emotional Approach Coping Scales | Change from baseline to 8 weeks
  Sum of eight self-report items assessing whether the subject uses an emotional approach to coping when experiencing stress or difficulties. Items range from 1-4 (1 = I don't use this emotional coping strategy; 4 = I use this emotional coping strategy a lot), yielding a total score between 8 and 32.
Emotional Approach Coping Scales | Change from baseline to 20 weeks
  Sum of eight self-report items assessing whether the subject uses an emotional approach to coping when experiencing stress or difficulties. Items range from 1-4 (1 = I don't use this emotional coping strategy; 4 = I use this emotional coping strategy a lot), yielding a total score between 8 and 32.
Pain Catastrophizing Scale | Change from baseline to 8 weeks
  Sum of thirteen self-report items assessing the types of thoughts and feelings experienced with pain. Items range from 0-4 (0 = not experiencing a type of thought / feeling; 5 = experiencing that thought / feeling all the time), yielding a total score between 0 and 52. Higher scores indicate the subject experiences thoughts and emotions that typically catastrophizes their pain.
Pain Catastrophizing Scale | Change from baseline to 20 weeks
  Sum of thirteen self-report items assessing the types of thoughts and feelings experienced with pain. Items range from 0-4 (0 = not experiencing a type of thought / feeling; 5 = experiencing that thought / feeling all the time), yielding a total score between 0 and 52. Higher scores indicate the subject experiences thoughts and emotions that typically catastrophizes their pain.
Survey of Pain Attitudes | Change from baseline to 8 weeks
  Sum of fourteen self-report items assessing the subject's attitude towards their pain. Items range from 0-4 (0 = this attitude is very untrue for me; 4 = this attitude is very true for me), yielding a total score between 0 and 56.
Survey of Pain Attitudes | Change from baseline to 20 weeks
  Sum of fourteen self-report items assessing the subject's attitude towards their pain. Items range from 0-4, yielding a total score between 0 and 56.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided